CLINICAL TRIAL: NCT04725058
Title: Obesity Group Visits. A Novel Way to Approach the Obesity Epidemic in an Inner-City Setting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Theodore Friedman, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1443169
Record Dates: First submitted 2021-01-11; First posted 2021-01-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Group Visit (Experimental): Participants receive obesity management in a group setting let by endocrinologist and nutritionist.
  Interventions: Other: Medical Group Visit
- Dietitian-Led Visit (Experimental): Participant receives obesity management in an individual setting lead by registered dietitian.
  Interventions: Other: Dietitian Individual Visit

INTERVENTIONS:
Other: Medical Group Visit — A group of 20 or more participants will receive obesity management through endocrinologist and registered dietitian in a group seetting.
  Other Names: Medical Group
  Arms: Medical Group Visit
Other: Dietitian Individual Visit — Participant receives obesity management individually from a registered dietitian.
  Arms: Dietitian-Led Visit

SUMMARY:
The purpose of this study has two aims: Aim 1: To compare a medical group visit model versus a dietitian-let model (shared composite group visit approach vs individualized dietitian-led approach) to provide obesity care in a real-world diverse inner city population.

Aim 2. To use both perivascular fat attenuation and coronary artery calcium (CAC) scores in those receiving composite group intervention vs. dietitian-led intervention to see if lifestyle intervention can reduce plaque progression and improve perivascular fat attenuation.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all study participants giving written informed consent will be screened to determine eligibility for study entry. At week 0, study participants who meet the eligibility requirements will be randomized in a blind manner (participant only) in a 3:1 block ratio. The study will randomize 750 subjects to the composite group visit and 250 subjects to the dietitian-led group into a 12-months duration study.

For Aim 2: A subset of 200 participants who identify as female and over 50 years old and males over 40 years old randomized to either the composite group arm or the dietitian-led arm will have the option to take part in a sub-study that involves getting a Coronary Artery Calcium (CAC) scan done at the Lundquist Institute. The first 125 subjects in the composite group arm and the first 75 subjects in the dietitian-led arm that express interest and want to undergo CAC scanning and perivascular fat measurements at baseline and at 12-months of intervention will need to sign a separate consent for these procedures. CAC scan readers will be blind to the assigned group. A group of 100 subjects not participating in the aim 1 intervention will be able to join the study under the control group. These participants will not be randomly assigned.

ELIGIBILITY:
* Inclusion

  * Age ≥ 18
  * BMI ≥ 30 kg/m2
  * Male, Female, LGBT
  * Any ethnicity
  * Interested in weight loss and be open to being randomized in either a medical group visit arm or dietitian-led arm (willingly agree to sign consent form)
  * Currently within or be eligible to receive care at LAC-DHS and be empaneled to have a primary care provider (PCP) who can adjust their medicines including anti-hypertensive and diabetic medications if needed.
  * If had stopped taking weight loss medication (orlistat, lorcaserin, and phentermine/topiramate-ER, phenetermine, diethylpropion, phendimetrazine and benzphetamine) for at least 2 months prior enrollment
  * If had stopped taking supplements advertised to increase weight loss at least 3 months prior enrollment

Females >50 years of age and Males >40 years of age meet inclusion criteria to participate in the sub-study that involves getting a Coronary Artery Calcium (CAC) scan done at the Lundquist Institute.

Exclusion Criteria:

* Age <18
* BMI< 30 kg/m2
* Unwilling to sing consent form
* Currently participating in another obesity treatment program
* Currently on a weight loss medication (orlistat, lorcaserin, and phentermine/topiramate-ER, phenetermine, diethylpropion, phendimetrazine and benzphetamine)
* Currently on metformin or topiramate primarily prescribed for weight loss
* Currently pregnant
* Ineligible to receive care at LAC-DHS
* Those with mental illness, substance abuse issues as well as other illnesses who are unable to follow directions related to the study or becomes disruptive to the overall group
* Patients who have had bariatric surgery less than a year from time of enrollment

Females <50 years of age and Males <40 years of age are not eligible to participate in the sub-study that involves getting a Coronary Artery Calcium (CAC) scan done at the Lundquist Institute.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | Baseline, months 3, 6 and 12.
  Weight will be measured at baseline and at 3,6, and 12 months.
Change in HbA1c | Baseline, months 3, 6 and 12.
  Hemoglobin A1c will be measured at baseline, and at moths 0, 3, 6 and 12 to determine the effect of the intervention arm.
Change in Healthy Eating Index-2015 Score | Baseline, months 3, 6 and 12.
  Diet quality will be assessed by the healthy eating Index-2015 score calculated from the food frequency questionnaire using the diet history questionnaire tool (DHQ) version III software. The minimum and maximum scores ranges fron 0 to 100. Higher scores greater than 60 indicate better diet quality.
Change in Physical Activity Measures | Baseline, months 3, 6 and 12.
  The IPAQ short form is a seven-item instrument evaluation tool of physical activity among the adults that measures a range of physical activity from vigorous to sedentary over the last 7 days. The specific type of activities assessed are walking, moderate intensity activities and vigorous intensity activities. All continuous scores are expressed in metabolic equivalent minutes(MET-minutes) per week with walking =3.3 METs, Moderate PA=4.0 METs and Vigorous PA = 8.0 METs. An overall total physical activity score can be computed as the sum of the total MET-minutes/week scores where more MET-minutes per week indicate more physical activity
Change in General Health Questionnaire (GHQ-12) Score | Baseline, months 3, 6 and 12.
  The General Health Questionnaire (GHQ-12) consists of 12-item rating scale for assessing psychological distress over the past few weeks. Scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress.
Change in Social Determinants of Health Factors (SDOH, PRAPARE (Protocol for Responding to and Addressing Patient Assets, Risks, and Experiences) tool. | Baseline and at month-12.
  Change from baseline to 12-month follow-up PRAPARE score. The PRAPARE assessment tool will be used to calculate a tally risk score indicating the cumulative number of SDOH risks a patient faces (including 15 SDOH domains).

SECONDARY OUTCOMES:
Change in Coronary Artery Calcification (CAC) score | Baseline and 12 months.
  Coronary Artery Scanning will be measured at baseline and at month 12 to determine calcium scores. The minimum and maximum scores ranges from 0 to 400. Higher scores means worse outcome. We categorized the total CAC scores into 0-100 no/mild risk; scores 101-400 moderate risk; and > 400 severe risk.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Friedman, MD. PhD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles R. Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: starting 6 months after publication.
Access Criteria: Contact Petra Duran and PI directly.

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Ryan DH, Bray GA. Pharmacologic treatment options for obesity: what is old is new again. Curr Hypertens Rep. 2013 Jun;15(3):182-9. doi: 10.1007/s11906-013-0343-6. PMID 23625271
- [Background] Carvajal R, Wadden TA, Tsai AG, Peck K, Moran CH. Managing obesity in primary care practice: a narrative review. Ann N Y Acad Sci. 2013 Apr;1281(1):191-206. doi: 10.1111/nyas.12004. Epub 2013 Jan 16. PMID 23323827
- [Background] Vadheim LM, Brewer KA, Kassner DR, Vanderwood KK, Hall TO, Butcher MK, Helgerson SD, Harwell TS. Effectiveness of a lifestyle intervention program among persons at high risk for cardiovascular disease and diabetes in a rural community. J Rural Health. 2010 Summer;26(3):266-72. doi: 10.1111/j.1748-0361.2010.00288.x. PMID 20633095